CLINICAL TRIAL: NCT01753115
Title: A Study of The Effects of Co-Administering Ciprofloxacin and BioThrax on the Pharmacokinetics of Ciprofloxacin in Healthy Adults
Brief Title: Ciprofloxacin BioThrax Co-Administration Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EBS.AVA.009
Record Dates: First submitted 2012-12-14; First posted 2012-12-20 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Anthrax
Keywords: post-exposure prophylaxis; toxin neutralization assay
MeSH Terms: conditions — Anthrax | interventions — Biothrax; Anthrax Vaccines; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BioThrax + Ciprofloxacin PK (Experimental): BioThrax: route of administration/schedule- 0.5 mL subcutaneous (SC) injection / 0-2-4 week schedule.
  Ciprofloxacin: 500 mg twice a day (Days 1-6, 19-21, 33-35, 40-48).
  Interventions: Biological: BioThrax; Drug: Ciprofloxacin
- BioThrax + Ciprofloxacin no PK (Experimental): BioThrax: route of administration/schedule- 0.5 mL subcutaneous (SC) injection / 0-2-4 week schedule.
  Ciprofloxacin: 500 mg twice a day (Days 1-6, 19-21, 33-35, 40-48).
  Interventions: Biological: BioThrax; Drug: Ciprofloxacin
- BioThrax only (Experimental): BioThrax: route of administration/schedule- 0.5 mL subcutaneous (SC) injection / 0-2-4 week schedule.
  Interventions: Biological: BioThrax

INTERVENTIONS:
Biological: BioThrax — route of administration/schedule- 0.5 mL subcutaneous (SC) injection / 0-2-4 week schedule
  Other Names: Anthrax Vaccine Adsorbed; AVA
Drug: Ciprofloxacin — 500 mg twice a day (Days 1-6, 19-21, 33-35, 40-48).
  Arms: BioThrax + Ciprofloxacin PK; BioThrax + Ciprofloxacin no PK

SUMMARY:
The purpose of this clinical trial is to determine whether there is any effect on the antibiotic, ciprofloxacin when taken before and after administration of a 3-dose series of BioThrax® (Anthrax Vaccine Adsorbed or AVA).

This study will be conducted in the United States (US) in 154 healthy male and female volunteer subjects ages 18 to 45.

The duration of study participation for each subject will be approximately 76 days (approximately 2.5 months)

DETAILED DESCRIPTION:
BioThrax is the only FDA-licensed vaccine for the prevention of anthrax infection. This is a randomized, open-label, Phase 2, multi-center trial to investigate the potential interactions of ciprofloxacin and BioThrax.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 45 years of age, at the time of enrollment
* Be in good health as determined by the investigator from medical history and a physical examination.
* If a pre-menopausal female, must be using acceptable methods of birth control.
* Be willing and able to return for all follow-up visits and blood and urine collections for the duration of the trial
* Be willing and able to complete a web-enabled electronic diary and report concomitant medications, adverse events, and BioThrax reactogenicity events during the trial
* Be able to understand and communicate in English.

Exclusion Criteria:

* Prior immunization with anthrax vaccine or known exposure to anthrax organisms
* Intend to enlist in the military during the study.
* Have a known allergy to aluminum hydroxide, formaldehyde, benzethonium chloride, or latex.
* Plan to receive experimental products 30 days prior to study entry or at any time during the study
* Have received a live vaccine in the 30 days before study entry
* Plan to receive a live vaccine at any time during the study.
* Have ongoing drug abuse/dependence (including alcohol) issues and/or test positive in a urine drug screen for amphetamines, barbiturates, cocaine or opiates
* Have received immunosuppressive therapy (including systemic steroids) within 30 days prior to trial entry
* Have any other condition known to produce or be associated with immunosuppression
* Have received cytotoxic therapy in the previous 5 years
* A chronic condition that, in the opinion of the Investigator, would render vaccination unsafe or would interfere with trial evaluations or completion of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hopkins, MD, MPH, TM, Principal Investigator — Emergent BioSolutions Inc.
Locations (3):
- United States (3):
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Meridian Clinical Research, Omaha, Nebraska
  - Research Across America, Dallas, Texas

REFERENCES:
- [Result] Cassie D, Longstreth J, Hopkins R, Hunter-Stitt E, Drobic B, Bellani M. Compatible co-administration of BioThrax(R) vaccine and ciprofloxacin-Results of a randomized open-label drug-vaccine interaction trial. Vaccine X. 2024 Jan 7;17:100431. doi: 10.1016/j.jvacx.2024.100431. eCollection 2024 Mar. PMID 38352727

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 14 Dec 2012 to 04 Aug 2013 at 3 US sites.
Groups:
- BioThrax + Ciprofloxacin PK; BioThrax + Ciprofloxacin no PK: BioThrax: route of administration/schedule- 0.5 mL subcutaneous (SC) injection / 0-2-4 week schedule
  Ciprofloxacin: 500 mg twice a day
Period: Overall Study
Arm/Group | BioThrax + Ciprofloxacin PK | BioThrax + Ciprofloxacin no PK | BioThrax Only
Started | 44 | 40 | 70
Treated | 38 | 39 | 67
Completed | 32 | 25 | 56
Not Completed | 12 | 15 | 14
Not completed — Lost to Follow-up | 3 | 6 | 8
Not completed — Withdrawal by Subject | 6 | 5 | 6
Not completed — Subject non-compliant | 3 | 3 | 0
Not completed — Used excluded drug | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat population: all subjects who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | BioThrax + Ciprofloxacin PK | BioThrax + Ciprofloxacin no PK | BioThrax Only | Total
Number analyzed (Participants) | 44 | 40 | 70 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (8.76) | 30.8 (8.05) | 30.2 (7.29) | 30.4 (7.88)
Age, Customized [Number; unit: participants]
  18 - 30 years | 22 | 20 | 35 | 77
  31 - 45 years | 22 | 20 | 35 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 36 | 76
  Male | 24 | 20 | 34 | 78
Race/Ethnicity, Customized [Number; unit: participants]
  White | 24 | 22 | 33 | 79
  Black or African America | 20 | 14 | 34 | 68
  Asian | 0 | 2 | 1 | 3
  American Indian or Alaskan Native | 0 | 1 | 2 | 3
  Multiple | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Ratios of Ciprofloxacin Area Under the Curve and Cmax (Day 5/Day 44)
Description: Ratios of Area Under the Curve from zero to 12 hours (AUC0-12h) and maximum concentration (Cmax) achieved for ciprofloxacin (Day 5/Day 44).
Time Frame: Day 5 and Day 44 in Arm 1
Population: Per protocol population: all subjects in arm 1 who received any dose of ciprofloxacin, had adequate PK data on Day 5 and Day 44, had received all three BioThrax doses, and who had no key protocol deviations (e.g., insufficient blood sample) that would be expected to affect the ciprofloxacin PK assessment.
Measure: Mean (90% Confidence Interval); unit: ratio
Groups:
- Arm 1 = BioThrax (0.5 mL) + Ciprofloxacin (500 mg Bid) + PK: BioThrax: route of administration/schedule- 0.5 mL subcutaneous (SC) injection / 0-2-4 week schedule
  Ciprofloxacin: 500 mg twice a day
Arm/Group | Arm 1 = BioThrax (0.5 mL) + Ciprofloxacin (500 mg Bid) + PK
Number analyzed (Participants) | 32
ratio
  Ratio Cmax Day 44/Day 5 | 0.944 [0.852 to 1.046]
  Ratio AUC0-12hr Day 44/Day 5 | 0.887 [0.831 to 0.948]
Statistical Analysis 1: Comparison: Arm 1 = BioThrax (0.5 mL) + Ciprofloxacin (500 mg Bid) + PK; Analysis of Ciprofloxacin Area Under the Curve at Day 5 and Day 44; Test type: Non-Inferiority or Equivalence — Equivalence margin is 0.80 - 1.25; Ratio of AUC = 0.887, 90% CI 2-sided [0.831 to 0.948]
Statistical Analysis 2: Comparison: Arm 1 = BioThrax (0.5 mL) + Ciprofloxacin (500 mg Bid) + PK; Analysis of Cmax at Day 5 and Day 44; Test type: Non-Inferiority or Equivalence — Equivalence margin is 0.80 - 1.25; Ratio of Cmax = 0.944, 90% CI 2-sided [0.852 to 1.046]

2. Secondary Outcome: Geometric Mean Titer (GMT) of Toxin Neutralizing Antibody (TNA) Levels
Description: Blood was collected in arms 1 and 2 at day 48 ( 2 weeks following last vaccination) and in arm 3 at day 43 ( 2 weeks following last vaccination) for TNA assay to determine the NF50 antibody titer for calculating GMT.
Time Frame: Two weeks after last vaccination
Population: BioThrax immunogenicity population: received 3 vaccinations and had samples taken within the study-specified windows; had a valid immunogenicity result within 2 wks of the last vaccination; had no evidence of previous anthrax vaccination and received the correct BioThrax dose at all 3 times; received vaccine maintained at the proper temperature.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- BioThrax + Ciprofloxacin (Arms 1 + 2): BioThrax: route of administration/schedule- 0.5 mL subcutaneous (SC) injection / 0-2-4 week schedule
  Ciprofloxacin: 500 mg twice a day
- BioThrax Only (Arm 3): BioThrax: route of administration/schedule- 0.5 mL subcutaneous (SC) injection / 0-2-4 week schedule
Arm/Group | BioThrax + Ciprofloxacin (Arms 1 + 2) | BioThrax Only (Arm 3)
Number analyzed (Participants) | 50 | 50
titer | 1.170 [0.912 to 1.500] | 0.923 [0.723 to 1.780]
Statistical Analysis 1: Comparison: BioThrax + Ciprofloxacin (Arms 1 + 2) vs BioThrax Only (Arm 3); Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.67; Ratio of GMT = 1.267, 95% CI 2-sided [0.898 to 1.787]

ADVERSE EVENTS:
Time Frame: Arm 1: enrollment, Days 0-5, 20, 34, 39-44, 48, or the early withdrawal visit (EWV) for a max of 16 visits. Arm 2: enrollment, Days 1, 5, 20, 34, 48, or EWV for a max of 6 visits. Arm 3: enrollment, Days 1, 15, 29, 43, or EWV for a max of 5 visits.
Description: Subjects in the safety (treated) population were asked about adverse event (AEs) at each visit. Severe (Grade 3) injection site and systemic reactions recorded in subject diaries were also recorded as AEs in the eCRF. Abnormal lab results, vital signs, and physical examination findings considered clinically significant were also recorded as AEs.
Arm/Group | BioThrax + Ciprofloxacin PK | BioThrax + Ciprofloxacin no PK | BioThrax Only
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/39 | 0/67
Other Adverse Events (participants affected / at risk) | 6/38 | 7/39 | 14/67
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BioThrax + Ciprofloxacin PK (N=38) | BioThrax + Ciprofloxacin no PK (N=39) | BioThrax Only (N=67)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 5 (9)
Fatigue (General disorders) | 0 (0) | 2 (4) | 3 (4)
Injection site erythema (General disorders) | 2 (2) | 0 (0) | 2 (3)
Injection site mass (General disorders) | 0 (0) | 0 (0) | 4 (5)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 4 (6)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (6)
Headache (Nervous system disorders) | 3 (3) | 4 (4) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor is responsible for public disclosure of study data. Any proposed publication is subject to review agreed between the Biomedical Advanced Research & Development Authority (BARDA) and Emergent; between Emergent and the contract research organizations (CROs)/vendors; and between the CROs and the site Principal Investigator. Data are the property of the sponsor and cannot be published without prior authorization from the sponsor, but data and publication thereof will not be unduly withheld.